CLINICAL TRIAL: NCT06831279
Title: Comparison of Two Different Rehabilitation Approaches Applied After Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MarmaraU- AYDOĞDU- ÜNAL001
Record Dates: First submitted 2025-01-09; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-05

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Anterior Cruciate Ligament; physical therapy; Dual Task; Foam Roller; Balance Exercise
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXERCISE GROUP (Active Comparator)
  Interventions: Other: EXERCISE
- FOAM ROLLER GROUP (Experimental): Bu grupta ek olarak hamstring kas grubuna dinamik şekilde foam roller ile uygulama yapılmıştır.
  Interventions: Other: EXERCISE

INTERVENTIONS:
Other: EXERCISE — Conventional Physiotherapy + Dual-Task Approach During Walking and Balance Exercises:

SUMMARY:
The anterior cruciate ligament is incumbent upon the stabilization of the knee joint in our body. Consequently, it is also of great importance for athletes since it is seen that injuries in clinics are predominantly monitored in young individuals, who do active sports. Anterior cruciate ligament injuries commonly occur in football players when a secondary task (motor or cognitive) is involved while they are busy with a motor activity. In these processes, a circumstance, in which there becomes a quick landing after a jump or a difficult pass whilst dribbling the ball, can be monitored. In such cases, the subject of preventing these injuries, which may occur in athletes, and making them ready for second tasks after the treatment of the injury, has become a current issue. It is important for individuals who have suffered the injury- to be able to bring the knee joint to its former function at the highest level after anterior cruciate ligament reconstruction. As a result, the development of novel rehabilitation strategies has been an ongoing focus of research. A prime exemplar of this phenomenon is the implementation of dual-task exercises. Dual-task exercises appear in athletes as motor-cognitive or motor-motor. Athletes' exercising motor-cognitive functions has attracted the attention of researchers in the past period to prevent injuries in sports and has brought a new breath to the academic world. Studies suggest a decrease in cognitive and motor functions in the acute period after injuries. However, observing its long-term effects, they also suggest an increase in the attention parameter, crucial for athletes.

In a study examining postural stability in individuals, who underwent an operation of anterior cruciate ligament reconstruction by giving motor-motor or motor-cognitive exercises, it is seen that worse results are obtained in postural stability in individuals, who underwent only anterior cruciate ligament reconstruction compared to healthy individuals. Furthermore, in cases -in which eyes were closed and dual motor tasks were given-, more negative results are obtained compared to the open-eyed group. It is associated with a significant decrease in proprioceptive performance in individuals after anterior cruciate ligament injury. Owing to this decrease, postural control decreases, and negative situations arise due to the pathology of the individual. The star balance test is a sensitive test to determine and emerges as an exercise that will correct this negative situation. Post-ACL injury, individuals exhibit significantly lower physical component scores in quality-of-life assessments compared to healthy controls, as reported in books and articles. Moreover, after the ACL reconstruction, a decrease in the mental scores of the individual is seen owing to reasons such as long-term absenteeism from work, rehabilitation, the high costs of the operation, and traumatic occasions.

Foam roller, one of the current treatment modalities, is a myofascial release technique. The purpose of the foam roller application is to activate myofascial release by using the athlete's body weight and back-and-forth movement cycle. It has been observed that the usage of foam roller delays the emergence of delayed muscle soreness with myofascial release in the quadriceps and hamstring muscles, while also increasing joint range of motion. Despite the widespread utilization of foam rollers in clinical practice, empirical evidence elucidating the underlying mechanisms and clinical efficacy of this modality remains relatively limited. Nevertheless, the factors -which are consequential in the return to pre-injury performance of the athletes- have not been thoroughly scrutinized. For instance, there is no encounter in the literature examining the effects of dual-task exercises on kinesiophobia, ACL-specific quality of life, star balance test evaluation, normal range of motion evaluation, Tegner-Lysholm knee scoring scale.

The purpose of the study is to compare two different rehabilitation groups in terms of pain, range of motion, functionality, balance, quality of life, and kinesiophobia in individuals who underwent ACL reconstruction. The first group is the one with a dual-task approach given during walking and balance exercises together with the conventional physiotherapy program. The latter is the one with the same dual-task approach given during walking and balance exercises together, as an extra with a foam roller.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing anterior cruciate ligament (ACL) reconstruction. Use of hamstring tendon autograft. Age between 18 and 40 years. At least 1 week but no more than 1 year post-surgery.

Exclusion Criteria:

* Presence of cardiovascular diseases. Any additional lower extremity disability (e.g., revision ACL reconstruction, other knee surgeries).

Diagnosis of back or lumbar pain. Any neurological disorders that could affect balance (e.g., epilepsy). Presence of posterior cruciate ligament (PCL) tear in addition to ACL injury.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Star Excursion Balance Test | At the baseline
  Dynamic balance was measured using the Yıldız Balance Test (YBT). Athletes will reach with their feet to the directions of a star drawn on the ground with a 45° angle, resulting in a total of 8 directions. The distance they can reach will be recorded in centimeters.
  Prior to the test, athletes will be given 3 minutes to familiarize themselves with the test, and there will be a 2-minute rest between trials. Additionally, a 5-second period will be allowed for the athletes to stand on both feet between each reach. The balance score is calculated using the formula "distance/leg length x 100" (Sitti S., 2013). If a volunteer cannot maintain balance on one foot, falls, pulls their hands away from their waist, or feels pain, the test is terminated.
Star Excursion Balance Test | Eight week later
  Dynamic balance was measured using the Yıldız Balance Test (YBT). Athletes will reach with their feet to the directions of a star drawn on the ground with a 45° angle, resulting in a total of 8 directions. The distance they can reach will be recorded in centimeters.
  Prior to the test, athletes will be given 3 minutes to familiarize themselves with the test, and there will be a 2-minute rest between trials. Additionally, a 5-second period will be allowed for the athletes to stand on both feet between each reach. The balance score is calculated using the formula "distance/leg length x 100" (Sitti S., 2013). If a volunteer cannot maintain balance on one foot, falls, pulls their hands away from their waist, or feels pain, the test is terminated.

SECONDARY OUTCOMES:
Quality of Life Assessment: (ACL-QOL Questionnaire) | At the baseline
  ACL-QOL is the only valid and reliable scale that measures the quality of life from the patient's perspective, rather than clinical criteria specific to ACL injuries, and it is available in Turkish. (Kinikli GI., 2015). This test examines 5 main areas with a total of 31 questions: symptoms and physical complaints (4 questions), work-related concerns (4 questions), hobbies, sports, or participation in competitions (12 questions), lifestyle (6 questions), and social and emotional aspects (5 questions).
Quality of Life Assessment: (ACL-QOL Questionnaire) | Eight week later
  ACL-QOL is the only valid and reliable scale that measures the quality of life from the patient's perspective, rather than clinical criteria specific to ACL injuries, and it is available in Turkish. (Kinikli GI., 2015). This test examines 5 main areas with a total of 31 questions: symptoms and physical complaints (4 questions), work-related concerns (4 questions), hobbies, sports, or participation in competitions (12 questions), lifestyle (6 questions), and social and emotional aspects (5 questions).
Tegner and Lysholm Rating Systems | At the baseline
  The Lysholm score was first investigated and developed in the 1970s. The Lysholm rating system is a 100-point scale consisting of 8 different items, with questions specifically related to instability and pain. It has been validated and is reliable in Turkish. (Çelik D., 2013). The Tegner activity score is a system with a scoring range of 0-10, including questions about daily life and sports activities. (Briggs KK., 2006).
Tegner and Lysholm Rating Systems | Eight week later
  The Lysholm score was first investigated and developed in the 1970s. The Lysholm rating system is a 100-point scale consisting of 8 different items, with questions specifically related to instability and pain. It has been validated and is reliable in Turkish. (Çelik D., 2013). The Tegner activity score is a system with a scoring range of 0-10, including questions about daily life and sports activities. (Briggs KK., 2006).
Range of Motion | At the baseline
  The normal range of motion for the knee joint is measured by moving the joint from the starting position of a typical universal goniometer to the end position of the entire range of motion, and recording the number indicated on the goniometer. In this study, a universal goniometer will be used to measure knee joint range of motion for both flexion and extension.
Range of Motion | Eight week later
  The normal range of motion for the knee joint is measured by moving the joint from the starting position of a typical universal goniometer to the end position of the entire range of motion, and recording the number indicated on the goniometer. In this study, a universal goniometer will be used to measure knee joint range of motion for both flexion and extension.
Pain Scale | At the baseline
  Visual Analog Scales (VAS) are psychometric measurement tools that make it possible to quantify the intensity of a symptom as subjectively experienced by individuals. (Klimek, 2017). For pain assessment, a 100 mm paper is provided. One end of the paper is labeled 'no pain - 0' and the other end is labeled 'worst possible pain - 100'. The patient should mark the line according to their condition at the time of the assessment. (Myles et al., 2017). The point where the mark is placed is noted and recorded.
Pain Scale | Eight week later
  Visual Analog Scales (VAS) are psychometric measurement tools that make it possible to quantify the intensity of a symptom as subjectively experienced by individuals. (Klimek, 2017). For pain assessment, a 100 mm paper is provided. One end of the paper is labeled 'no pain - 0' and the other end is labeled 'worst possible pain - 100'. The patient should mark the line according to their condition at the time of the assessment. (Myles et al., 2017). The point where the mark is placed is noted and recorded.
Tampa Scale for Kinesiophobia (TSK): | At the baseline
  Kinesiophobia (fear of movement) was first introduced in 1990 and will be assessed using the Tampa Scale for Kinesiophobia (TSK). (Miller et al., 1991). The TSK is a questionnaire consisting of 17 items designed to assess the fear of re-injury due to a previous trauma. The primary questions address variables related to re-injury, fear, and avoidance of movement in relation to the person's occupation or activities. The TSK uses a Likert scale with 1, 2, 3, and 4 points (1: Strongly Disagree, 4: Strongly Agree). Scores range from 17 to 68. (Huang et al., 2019). A higher score on the scale indicates a higher level of fear of movement. (Demirbuken et al., 2016).

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided